CLINICAL TRIAL: NCT03937934
Title: Study Title: Food Rx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Erin C. Westfall, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-006630
Record Dates: First submitted 2019-04-30; First posted 2019-05-06 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Diabetes; High Blood Pressure; Obesity; Hypertension; Heart Diseases; Stroke; TIA; Osteoarthritis; Cancer
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Obesity; Heart Diseases; Stroke; Osteoarthritis; Neoplasms | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with long term health condition (Experimental): Subjects that have been identified as having food insecurity based on a two question screening tool, and also has one of more of the following chronic diseases Hypertension, Heart disease, Stroke/TIA, DM 2, Cancer/history of cancer, obesity or osteoarthritis will receive weekly nutrition educaiton
  Interventions: Behavioral: Nutrition Education

INTERVENTIONS:
Behavioral: Nutrition Education — Weekly box of healthy groceries and nutrition education including a recipe, food to make the recipe, extra fruit and vegetables.

SUMMARY:
Researchers are trying to determine if subjects with lack of access to healthy food and a long term health problem, are helped by a weekly box of healthy groceries and nutrition education.

DETAILED DESCRIPTION:
Participants that have a chronic preventable disease and food insecurity will be offered enrollment in the study. Once all participants are enrolled, they will be given weekly boxes of food which includes materials for a nutritious recipe and extra fruit and vegetables for a total of 6 weeks. The SNAP-Ed Educator and SHIP Public health coordinator will be present at food pick up to answer questions about the boxes, food preparation, etc. They will be given the option of participating in grocery store and farmer's market tours, as well as sign up for text messaging of nutrition information and recipes. At the end of 6 weeks, they will be asked to participate in a focus group. At baseline, 3 months and 6 months, they will be asked to complete a survey on lifestyle behaviors and food choices.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients that have been identified as having food insecurity based on a two question screening tool, AND
* Also has one of more of the following chronic diseases:
* Hypertension,
* Heart disease,
* Stroke/TIA,
* DM 2,
* Cancer/history of cancer,
* obesity
* osteoarthritis

Exclusion Criteria:

* Pregnant women
* Children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Change in the number of self-reported fruits per day | Baseline, 3 months, 6 months
  Number of self-reported fruits per day
Change in the number of self-reported vegetables per day | Baseline, 3 months, 6 months
  Number of self-reported vegetables per day
Change in number of days a week and minutes per day participants participate in physical activity and sedentary activity | Baseline, 3 months, 6 months
  Measured using self-reported Food Rx Pilot survey

SECONDARY OUTCOMES:
Change in A1c | 6 months and 12 months
  Identified through chart review
Change in BMI kg/m2 (weight in kg, height in meters) | 6 months and 12 months
  Identified through chart review
Change in Systolic and/or Diastolic Hypertension mmHg | 6 months and 12 months
  Identified through chart review

CONTACTS AND LOCATIONS:
Overall Officials: Erin Westfall, DO, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Health System, Mankato, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials